CLINICAL TRIAL: NCT02335866
Title: Platelet Rich Fibrin Against Connective Tissue Graft in Treatment of Gingival Recessions
Brief Title: Platelet-Rich Fibrin in the Treatment of Multiple Gingival Recessions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, ELİF ONCU, Assist.Prof.Dr., Necmettin Erbakan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/10
Record Dates: First submitted 2014-12-13; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Gingival Recessions
Keywords: Platelet rich fibrin; Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test groups. (Experimental): This clinical study was designed as a split-mouth, randomized, controlled clinical trial. Bilateral gingival recession defects were randomly assigned to the test (CAF+PRF) or the control (CAF+SCTG) groups with the use of computer-generated randomization table after assessment of clinical parameters at baseline.
  Interventions: Procedure: test groups
- Control groups. (Active Comparator): This clinical study was designed as a split-mouth, randomized, controlled clinical trial. Bilateral gingival recession defects were randomly assigned to the test (CAF+PRF) or the control (CAF+SCTG) groups with the use of computer-generated randomization table after assessment of clinical parameters at baseline.
  Interventions: Procedure: Control groups

INTERVENTIONS:
Procedure: test groups — At the test sites, the previously prepared PRF was positioned over the recession defects, the coronal margin of the PRF was placed at the CEJ
  Other Names: PRF groups
  Arms: Test groups.
Procedure: Control groups — Split-full-split thickness flap incisions were performed in a coronal-apical direction. The papillae adjacent to the involved tooth were de-epithelialized to create a connective tissue bed. The gingival flap was repositioned without tension, with its margin located on the enamel, on the test and control sides. It was held in that position with 5-0 resoble sutures
  Other Names: Connective tissue graft groups
  Arms: Control groups.

SUMMARY:
The main objective of this study was to evaluate the clinical effectiveness of platelet-rich fibrin membrane used in combination with a coronally advanced flap and to compare it with the use of a subepitelial connective tissue graft in combination with a coronally advanced flap in Miller class I-II bilateral gingival recession treatment

DETAILED DESCRIPTION:
Purpose

The main objective of this study was to evaluate the clinical effectiveness of platelet-rich fibrin (PRF) in combination with modified coronally advanced flap (MCAF) in the treatment of multiple gingival recessions. Furthermore the second aim of the present study was to compare plastic periodontal surgical procedure, with PRF membrane and connective tissue graft, by a randomized splitmouth controlled study.

Clinical effectiveness of platelet-rich fibrin (PRF) in combination with modified coronally advanced flap (MCAF) as measured by Clinical measurements.

Material and Methods

Twenty patients with multiple gingival recession defects (Miller I, II) participated in this split-mouth trial. Sixty defects received either MCAF+PRF (test) or MCAF with subepithelial connective tissue graft (SCTG) (control). Gingival recession depth (RD), gingival recession width (RW), keratinized tissue width (KTW), recession area (RA), probing depth (PD), clinical attachment level (CAL) and gingival thickness (GT) were evaluated at baseline and 6 months. Additionally post-surgery patient satisfaction and pain status were measured by comparing visual analogue scale (VAS) scores.

Clinical measurements were taken at starting point and 6 months postoperatively. The measurements comprised an assessment of probing depth (PD),clinical attachment level (CAL) and gingival recession parameters including recession depth (RD), recession width (RW), keratinized tissue width (KTW) and gingival thickness (GT) were assessed by a calibrated examiner (E. Ö.). PD, CAL, RD, RW and KTW values were recorded by a Williams probe graduated in 1-mm increments and rounded up to the nearest millimeter (Hu Friedy, Chicago, IL, USA). To standardize the clinical measurements acrylic stents were prepared on patients' casts. The following measurements were recorded at the mid-buccal point of the teeth at baseline and6 months after surgery. GT was evaluated using endodontic reamer attached to a rubber stopper inserted perpendicularly into the gingival tissue 3 mm below the gingival margin under local anesthesia, and then the thickness was measured to the nearest 0.1 mm using a caliper.RD was measured from the CEJ to the gingival margin, RW was measured tangentially at the mid-facial CEJ and RA was calculated as the area within the contour of denuded root. KTW recorded as the distance from the mucogingival junction to the gingival margin. Duplicate measurements were made for RD, RW, RA and KTW with an interval of 24 hours and the average value of two measurements was used for the assessment. The postoperative pain was evaluated with a visual analog score (VAS).

ELIGIBILITY:
Inclusion Criteria:

* non smoking,
* similar bilateral Miller Class I or II20 localized gingival recessions at least ≥3 mm, located on incisors, canines or premolars on both jaws,
* identifiable cemento-enamel junction (CEJ),
* age ≥18 years,
* presence of tooth vitality and absence of restorations and superficial caries in the area to be treated,
* no periodontal surgical treatment on the involved sites,
* sufficient palatal donor tissue at least ≥2.5 mm thickness for the indicated SCTG

Exclusion Criteria:

* Patients in a pregnancy or lactation period or with self-reported history of antibiotic medication within 6 months
* Molar, mobile or fully restorated teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Change from baseline in gingival recession will be assessed at 1, 3 and 6 months.
Gingival recession depth | 6 months
  Change from baseline in gingival recession will be assessed at 6 months

SECONDARY OUTCOMES:
Keratinized tissue width | 6 months
  Change from baseline in keratinized tissue at 6 months.
Pain scores | first week after operations
  Pain level evaluated on visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: ELİF ÖNCÜ, PhD, Study Director — NECMETTİN ERBAKAN UNIVERSITY
Locations (1):
- NEU Dental School, Konya, Turkey (Türkiye)